CLINICAL TRIAL: NCT03499444
Title: A Phase 1, Open-label, Safety and Pharmacokinetic Study of Rucaparib in Japanese Patients With a Previously-treated Solid Tumor
Brief Title: A Study of Rucaparib in Japanese Patients With a Previously-treated Solid Tumor
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: pharmaand GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CO-338-081
Record Dates: First submitted 2018-03-26; First posted 2018-04-17 (Actual); Last update posted 2023-06-09 (Actual); Status verified 2023-06

CONDITIONS: Advanced Solid Tumor
MeSH Terms: interventions — rucaparib

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Oral Rucaparib monotherapy (Experimental): Part I: Dose Escalation, Part II: Dose Expansion (Additional patients will be enrolled at the recommended dose as defined in Part I of the study.)
  Interventions: Drug: Rucaparib

INTERVENTIONS:
Drug: Rucaparib — Rucaparib will be administered twice daily
  Other Names: CO-338

SUMMARY:
This is a Phase 1 open-label, dose-escalation, safety and pharmacokinetic study of rucaparib administered twice daily (BID) to Japanese patients with a solid tumor who have failed previous standard treatment for their cancer. A recommended dose of rucaparib for Japanese patients will be determined in a dose-escalation portion and then further evaluated in a dose-expansion portion of the study.

ELIGIBILITY:
Inclusion Criteria:

* Be 20 years of age at the time the informed consent form is signed and of Japanese ethnicity (ie, both parents are native Japanese and were born in Japan).
* Have a solid tumor that has progressed on standard treatment:

  * For patients enrolled in the dose-escalation portion, has confirmed solid tumor that is locally recurrent or metastatic
  * For patients enrolled in the dose-expansion portion, has high-grade serous ovarian cancer, or BRCA 1/2 mutated breast cancer, or other solid tumor with BRCA 1/2 or related gene mutation
* Have to have evaluable disease (i.e. disease can be followed on scans.)
* Be willing and able to fast for at least 14 hours

Exclusion Criteria:

* Active second malignancy
* Prior treatment with any PARP inhibitor
* Symptomatic and/or untreated CNS metastases
* Women who are breastfeeding or pregnant
* Pre-existing duodenal stent and/or any gastrointestinal disorder that would interfere with drug absorption
* Requires regular blood transfusions

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2018-02-06 (Actual); Primary Completion 2019-06-18 (Actual); Study Completion 2022-04-13 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment-related Adverse Events (AEs) as assessed by CTCAE v4.03 as a measure of safety and tolerability | From enrollment to completion of Part I (up to 12 months)
Number of participants with serious AEs as a measure of safety and tolerability | From enrollment to completion of Part I (up to 12 months)
Number of participants with worsening laboratory values as a measure of safety and tolerability | From enrollment to completion of Part I (up to 12 months)

SECONDARY OUTCOMES:
Dose-limiting toxicities (DLTs) during Cycle 1 of treatment | From enrollment to completion of Part I (up to 12 months)
Area under the plasma concentration versus time curve [AUC] | From enrollment to completion of Part I (up to 12 months)
Peak Plasma Concentration [Cmax] | From enrollment to completion of Part I (up to 12 months)
Total Plasma Clearance [CI/F] | From enrollment to completion of Part I (up to 12 months)
Response to treatment according to RECIST Version 1.1 | From enrollment to primary completion of study (up to 3 years)

CONTACTS AND LOCATIONS:
Locations (3):
- Japan (3):
  - Division of Medical Oncology, Hyogo Cancer Center, Akashi, Hyōgo
  - Department of Gynecologic Oncology, Saitama Medical Univeristy international Medical Center, Hidaka, Saitama
  - Department of Breast and Medical Oncology, National Cancer Center Hospital, Tsukiji, Tokyo